CLINICAL TRIAL: NCT05284812
Title: A Phase Ⅱ Study on the Safety, Tolerability and Immunogenicity of the Recombinant Mycobacterium Tuberculosis Vaccine Freeze-dried
Brief Title: A Phase Ⅱ Clinical Trial of the Recombinant Mycobacterium Tuberculosis Vaccine Freeze-dried (AEC/BC02)
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: It is planned to restart the clinical study after the completion of the clinical trial protocol modification.
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LKM-2021-BJH01
Record Dates: First submitted 2022-02-21; First posted 2022-03-17 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Vaccine
MeSH Terms: conditions — Tuberculosis | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Negative control population group (No Intervention): In population I, 20 subjects were considered to be recombinant mycobacterium tuberculosis fusion protein (EC) and BCG pure protein derivative (BCG-PPD) skin test results were negative.The type I population did not take chemical drugs and was not vaccinated, and was only used as immunogenicity control.
- Sentinel group (Other): In Population Ⅱ, 20 subjects were considered to be recombinant mycobacterium tuberculosis fusion protein (EC) was positive. First, 5 people aged 18-59 years were selected for low dose injection, 5 people aged 18-59 years were selected for high dose injection, 5 people aged ≥60 years were selected for low dose injection, and 5 people aged ≥60 years were selected for high dose injection.The subjects received a total of 6 doses of the vaccine, 1 dose every 2 weeks.
  Interventions: Biological: Low-dose freeze-dried recombinant tuberculosis vaccine (AEC / BC02); Biological: High-dose freeze-dried recombinant tuberculosis vaccine (AEC / BC02)
- Low-dose group (Experimental): In population Ⅲ, 40 subjects were considered to be recombinant mycobacterium tuberculosis fusion protein (EC) was positive. The type Ⅲ population were injected Low-dose freeze-dried recombinant tuberculosis vaccine (AEC / BC02).The subjects received a total of 6 doses of the vaccine, 1 dose every 2 weeks.
  Interventions: Biological: Low-dose freeze-dried recombinant tuberculosis vaccine (AEC / BC02)
- High-dose group (Experimental): In population Ⅳ, 40 subjects were considered to be recombinant mycobacterium tuberculosis fusion protein (EC) was positive. The type Ⅳ population were injected High-dose freeze-dried recombinant tuberculosis vaccine (AEC / BC02).The subjects received a total of 6 doses of the vaccine, 1 dose every 2 weeks.
  Interventions: Biological: High-dose freeze-dried recombinant tuberculosis vaccine (AEC / BC02)
- 3 dose of High-dose group (Experimental): In population Ⅴ, 40 subjects were considered to be recombinant mycobacterium tuberculosis fusion protein (EC) was positive. The type Ⅴ population were injected 3 dose of High-dose freeze-dried recombinant tuberculosis vaccine (AEC / BC02) and 3 dose of Lyophilized recombinant tuberculosis vaccine (AEC / BC02) placebo.The first, third, and sixth doses of the subjects were High-dose freeze-dried recombinant tuberculosis vaccine (AEC / BC02), and the second, fourth, and fifth doses were Lyophilized recombinant tuberculosis vaccine (AEC / BC02) placebo. Each dose is 2 weeks apart.
  Interventions: Biological: High-dose freeze-dried recombinant tuberculosis vaccine (AEC / BC02); Biological: Lyophilized recombinant tuberculosis vaccine (AEC / BC02) placebo
- Placebo group (Placebo Comparator): In population Ⅵ, 20 subjects were considered to be recombinant mycobacterium tuberculosis fusion protein (EC) was positive. The type Ⅵ population were injected Lyophilized recombinant tuberculosis vaccine (AEC / BC02) placebo.The subjects received a total of 6 doses of the vaccine, 1 dose every 2 weeks.
  Interventions: Biological: Lyophilized recombinant tuberculosis vaccine (AEC / BC02) placebo
- Adjuvant group (Active Comparator): In population Ⅶ, 20 subjects were considered to be recombinant mycobacterium tuberculosis fusion protein (EC) was positive. The type Ⅶ population were injected High-dose adjuvant for freeze-dried recombinant tuberculosis vaccine (AEC / BC02).The subjects received a total of 6 doses of the vaccine, 1 dose every 2 weeks.
  Interventions: Biological: High-dose adjuvant for freeze-dried recombinant tuberculosis vaccine (AEC / BC02)

INTERVENTIONS:
Biological: Low-dose freeze-dried recombinant tuberculosis vaccine (AEC / BC02) — Subjects receive low-dose freeze-dried recombinant tuberculosis vaccine (AEC / BC02) injection into the deltoid muscle of the upper arm
  Arms: Low-dose group; Sentinel group
Biological: High-dose freeze-dried recombinant tuberculosis vaccine (AEC / BC02) — Subjects receive high-dose freeze-dried recombinant tuberculosis vaccine (AEC / BC02) injection into the deltoid muscle of the upper arm
  Arms: 3 dose of High-dose group; High-dose group; Sentinel group
Biological: High-dose adjuvant for freeze-dried recombinant tuberculosis vaccine (AEC / BC02) — Subjects receive high-dose adjuvant for freeze-dried recombinant tuberculosis vaccine (AEC / BC02) injection into the deltoid muscle of the upper arm
  Arms: Adjuvant group
Biological: Lyophilized recombinant tuberculosis vaccine (AEC / BC02) placebo — Subjects receive Lyophilized recombinant tuberculosis vaccine (AEC / BC02) placebo injection into the deltoid muscle of the upper arm
  Arms: 3 dose of High-dose group; Placebo group

SUMMARY:
The safety, tolerability and immunogenicity of lyophilized recombinant tuberculosis vaccine (AEC/BC02) were studied in a randomized, blind, controlled phase ⅱ A clinical study in patients 18 years and older with latent infection of Mycobacterium tuberculosis.Twenty patients with negative control group and 180 patients with latent mycobacterium tuberculosis infection were divided into sentinel group, placebo group, high-dose adjuvant group, low-dose vaccine group, high-dose vaccine group and high-dose vaccine group (three doses).During the test, each subject shall not change groups or receive drugs.The negative control group did not take chemical drugs and did not get vaccinated after enrollment, and was only used as immunogenicity control.The latent infection group was given orally Koch inhibitor chemical drugs (Ifu tablet or Ifu capsule) or placebo twice a week, and then received placebo, adjuvant or vaccine every two weeks (0-2-4-6-8-10 weeks), with a total of 6 doses injected intramuscular alternately in the left and right arms of the upper arm deltoid muscle.

ELIGIBILITY:
Inclusion Criteria:

1. The age is 18 years old and above, and the gender is not limited;
2. I agree to participate in this study and sign the informed consent;
3. I can complete the whole process of clinical research in accordance with the requirements of the clinical research program;
4. Vital signs (reference range of normal values of vital signs: systolic blood pressure <160 mmHg and diastolic blood pressure <100 mmHg (which can be controlled by taking medicine), pulse 60-100 beats/min, axillary temperature <37.3 ℃ in a quiet state), Physical examination results show no abnormality or abnormality without clinical significance;
5. Negative control population: the test results are EC- and PPD- (the average diameter of EC skin test induration and flush is less than 5mm, and the PPD skin test induration is less than 5mm), and the chest imaging is normal;
6. People with latent infection of Mycobacterium tuberculosis: the test result is EC+ (EC skin test induration or flush ≥5mm), and the chest imaging is normal;
7. Laboratory tests including blood routine, urine routine, blood biochemistry and other tests are all normal or have no clinical significance;
8. There is no abnormality in the electrocardiogram examination or the abnormality has no clinical significance;
9. Those who have no history of tuberculosis after medical history inquiry.

Exclusion Criteria:

1. Those who are currently diagnosed with tuberculosis or have a history of tuberculosis and/or tuberculosis treatment;
2. There are serious chronic diseases or the disease is in the advanced stage and cannot be controlled smoothly, such as diabetes and thyroid disease;
3. Currently suffering from or within 2 years of any of the following serious diseases, such as: advanced tumor, autoimmune disease, progressive atherosclerosis, acute exacerbation of chronic obstructive pulmonary disease, acute or progressive liver or kidney disease, congestive heart failure exhaustion, etc.;
4. Those with known or suspected (or high-risk) immune function impairments or abnormalities, such as those receiving systemic glucocorticoids, immunosuppressants or immunosuppressants within 3 months, and within 3 months Those who received protein preparations or blood products or plasma extracts outside the gastrointestinal tract;
5. Existing mental/neurological diseases or history of mental/neurological diseases: those with convulsions, epilepsy, encephalopathy, or family history of mental illness;
6. Those who currently suffer from biliary obstruction;
7. People with allergic constitution, such as those with a history of allergy to two or more drugs or foods; a history of severe allergy to any component of the test vaccine, such as: anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenia Purpura, dyspnea, angioedema, etc.; or a history of the above-mentioned serious side effects after using any vaccine or drug in the past; a history of allergy to isoniazid tablets, rifampicin and rifamycin antibiotics;
8. Patients with severe liver insufficiency, or patients with drug-induced hepatitis and acute liver disease caused by any cause;
9. Difficulty swallowing, active or clinically significant digestive system diseases, and affecting drug absorption;
10. Current patients with active viral hepatitis and/or HIV antibody positive for human immunodeficiency virus and/or current or past syphilis;
11. Women who are pregnant, breastfeeding, or have a positive urine pregnancy test during the screening period, or before vaccination, or who have childbearing plans during the study period;
12. Those who are vaccinated with inactivated vaccine within 14 days before oral administration of chemical drugs, and those who are vaccinated with live attenuated vaccine within 30 days;
13. Those who have participated in any other clinical research and used the investigational drug within 3 months before this clinical research;
14. Any other situation that the researcher believes may affect the evaluation of the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of adverse events after intramuscular injection | Up to 6 months after the sixth time injection
  The observation of adverse events mainly come from vital sign detection and laboratory examination (including blood routine/urine routine/blood biochemistry/electrocardiogram and chest X-ray), local reactions and systemic reactions after injection.

SECONDARY OUTCOMES:
Laboratory markers of immunity | Up to 3 months after the sixth time injection
  Changes in the levels of antigen-specific total IgG antibodies and IgG subclasses (IgG1 and IgG2).
Laboratory markers of immunity | Up to 3 months after the sixth time injection
  Changes in the levels of antigen-specific IFN-γ levels.
Laboratory markers of immunity | Up to 3 months after the sixth time injection
  The changes of the proportion of antigen-specific T cells in PBMCs.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Huang, Bachelor, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan, China

REFERENCES:
- [Background] Pulendran B, Ahmed R. Immunological mechanisms of vaccination. Nat Immunol. 2011 Jun;12(6):509-17. doi: 10.1038/ni.2039. PMID 21739679
- [Background] Chen L, Xu M, Wang ZY, Chen BW, Du WX, Su C, Shen XB, Zhao AH, Dong N, Wang YJ, Wang GZ. The development and preliminary evaluation of a new Mycobacterium tuberculosis vaccine comprising Ag85b, HspX and CFP-10:ESAT-6 fusion protein with CpG DNA and aluminum hydroxide adjuvants. FEMS Immunol Med Microbiol. 2010 Jun 1;59(1):42-52. doi: 10.1111/j.1574-695X.2010.00660.x. Epub 2010 Feb 17. PMID 20298499
- [Derived] Li J, Fu L, Guo X, Yang Y, Dong J, Wang G, Zhao A. Novel BC02 Compound Adjuvant Enhances Adaptive and Innate Immunity Induced by Recombinant Glycoprotein E of Varicella-Zoster Virus. Vaccines (Basel). 2022 Dec 15;10(12):2155. doi: 10.3390/vaccines10122155. PMID 36560565